CLINICAL TRIAL: NCT02509039
Title: A Phase 1, Multi-center, Open-label Dose-escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of CC-122 Administered Orally to Adult Japanese Subjects With Advanced Solid Tumors or Non-Hodgkin's Lymphoma
Brief Title: A Study of CC-122 to Assess the Safety and Tolerability in Japanese Patients With Advanced Solid Tumors and Non-Hodgkin's Lymphoma (NHL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Replaced it with another clinical trial.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-122-ST-002
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-04

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: CC-122; Phase1; solid tumor; non-Hodgkin's lymphom
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione

ARMS (1):
- CC-122 (Experimental): CC-122 is administered orally, on a 5 continuous days out of 7 days per week intermittent dosing schedule.
  Interventions: Drug: CC-122

INTERVENTIONS:
Drug: CC-122 — 5 continuous days out of 7 days per week intermittent dosing

SUMMARY:
To determine the safety and tolerability of CC-122 when administered orally to adult Japanese subjects with advanced solid tumors or Non-Hodgkin's Lymphoma (NHL) and to define the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).

DETAILED DESCRIPTION:
This is a phase 1, multicenter, open-label, dose-escalation study that will evaluate the safety, tolerability, (Pharmacokinetics) PK, and preliminary efficacy of CC-122 in Japanese subjects with advanced solid tumors or Non-Hodgkin's Lymphoma (NHL).

Subjects will receive ascending dose levels of CC-122 from Cycle 1 onwards to measure PK and to determine safety and tolerability.

An initial cohort of at least three subjects will be given CC-122 at a dose of 2.0 mg on an intermittent dosing schedule (5 continuous days out of 7 days per week) and 3-6 subjects will be enrolled in subsequent dose levels. Dose escalation for subsequent cohorts will proceed according to a standard dose escalation design (3+3 design) (Storer, 1989) to establish initial toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent document prior to any study-related assessments/procedures are conducted
2. 20 years or older, with histological or cytological confirmation of advanced solid tumors or Non-Hodgkin's Lymphoma (NHL), including those who have progressed on standard anticancer therapy or for whom no other conventional therapy exists
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2 for all tumors
4. Subjects must have the following laboratory values:

   ・Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
   * Hemoglobin (Hgb) ≥ 9 g/dL, drawn at least 7 days after the last RBC transfusion
   * Platelets (Plt) ≥ 100 x 109/L, drawn at least 7 days after the last platelet transfusion
   * Potassium within normal limits or correctable with supplements
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN) or ≤ 5.0 x ULN if liver tumors are present
   * Serum bilirubin ≤ 1.5 x ULN; subjects with serum bilirubin >1.5 x ULN and ≤ 2 x ULN may be enrolled if agreed to by the sponsor
   * Serum creatinine ≤ ULN or 24-hour clearance ≥ 50 mL/min
   * Negative serum pregnancy test in females of childbearing potential as per the CC-122 Pregnancy Prevention Rist Management Plan
5. Able to adhere to the study visit schedule and other protocol requirements
6. Must adhere to the Pregnancy Prevention Rist Management Plan

Exclusion Criteria:

1. Subjects with primary central nervous system (CNS) malignancies or symptomatic central nervous system metastases. Subjects with brain metastases that have been previously treated and are stable for 6 weeks are allowed
2. Known acute or chronic pancreatitis
3. Any peripheral neuropathy ≥ NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) Grade 2
4. Persistent diarrhea or malabsorption ≥ NCI CTCAE Grade 2, despite medical management
5. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   * Left Ventricular Ejection Fraction (LVEF) < 45% as determined by Multiple Gated Acquisition Scan (MUGA) scan or Echocardiogram (ECHO)
   * Complete left bundle branch, or bifascicular block

     * Congenital long QT syndrome
     * Persistent or uncontrolled ventricular arrhythmias or atrial fibrillation
     * QTcF > 460 msec on screening electrocardiogram (ECG) (mean of triplicate recordings)
     * Unstable angina pectoris or myocardial infarction ≤ 3 months prior to starting CC-122
     * Troponin-T value >0.4 ng/mL or Brain Natriuretic Peptide (BNP) >300 pg/mL Subjects with baseline troponin-T >ULN or BNP >100 pg/mL are eligible but must and optimization of cardioprotective therapy.
   * Other clinically significant heart disease such as congestive heart failure requiring treatment or uncontrolled hypertension (blood pressure ≥ 160/95 mmHg)
6. Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half lives or 4 weeks, whichever is shorter, prior to starting CC-122 or who have not recovered from side effects of such therapy. Luteinizing hormone-releasing hormone (LHRH) agonists will be allowed for subjects with metastatic prostate cancer
7. Major surgery ≤ 2 weeks prior to starting CC-122 or still recovering from post operative side effects
8. Women who are pregnant or breast feeding. Adults of reproductive potential not employing two forms of birth control as per Pregnancy Prevention Risk Management Plan (PPRMP)
9. Known human immunodeficiency virus (HIV) infection
10. Known acute or chronic hepatitis B or C virus infection
11. Status post solid organ transplant
12. Less than 100 days for subjects receiving autologous hematologic stem cell transplant (HSCT); or 6 months for subjects receiving allogeneic HSCT, or if otherwise not fully recovered from HSCT-related toxicity

    a. The 6-month exclusionary period for recovery from HSCT-associated toxicity, applies regardless of whether an autologous or allogeneic transplant was performed
13. Known hypersensitivity to any component of the formulation of CC-122
14. Any significant medical condition (including active or controlled infection or renal disease), laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
15. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
16. Any condition that confounds the ability to interpret data from the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- Japan (3):
  - Local Institution - 002, Koto-ku, Tokyo
  - Local Institution - 003, Chikusa-ku
  - Local Institution - 001, Kashiwa

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 participants treated
Groups:
- AIC 2.0 mg: CC-122 administered orally at a dose of 2.0 mg on a 5 continuous days out of 7 days per week intermittent dosing schedule using active ingredient in capsule (AIC)
- AIC 3.0 mg: CC-122 administered orally at a dose of 3.0 mg on a 5 continuous days out of 7 days per week intermittent dosing schedule using active ingredient in capsule (AIC)
- AIC 4.0 mg: CC-122 administered orally at a dose of 4.0 mg on a 5 continuous days out of 7 days per week intermittent dosing schedule using active ingredient in capsule (AIC)
- F6 3.0 mg: CC-122 administered orally at a dose of 3.0 mg on a 5 continuous days out of 7 days per week intermittent dosing schedule using formulated capsules (F6)
Period: Overall Study
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Started | 3 | 3 | 3 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 6
Not completed — Adverse Event | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Progressive disease | 2 | 2 | 1 | 5
Not completed — Study terminated by Sponsor | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (4.51) | 62 (14.53) | 68.7 (8.62) | 65.3 (7.5) | 64.6 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 3 | 6
  Male | 1 | 2 | 3 | 3 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Primary Race: Japanese | 3 | 3 | 3 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: NCI CTCAE Version 4.03 will be used to grade adverse events. Events described below will be classified as DLTs:
  * Non-hematologic AEs: Suspected to be related to CC-122, commences during the DLT evaluation period, and is ≥ Grade 3
  * Laboratory abnormalities: Suspected to be related to CC-122, commences during the DLT evaluation period, and is ≥ Grade 3
  * Hematologic: Any febrile neutropenia, Grade 4 neutropenia lasting > 7 days, Grade 4 thrombocytopenia lasting > 24 hours or thrombocytopenia of any grade requiring platelet transfusions, Any Grade 3/4 thrombocytopenia with clinically significant bleeding
  * Hepatic: Grade 4 liver function tests or Grade 3 ALT with Grade 2 or higher bilirubin will be considered a DLT, irrespective of underlying attribution. Other Grade 3 LFTs due to disease progression in the liver will not be considered DLTs
  * Other adverse events: Suspected to be related to CC-122 and necessitating a dose reduction during the DLT evaluation period
Time Frame: From first dose up to at least 28 days (Cycle 1)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD is defined as the last dose level below the non-tolerated dose (NTD) with zero or one out of six evaluable participants experiencing dose-limiting toxicities (DLTs) during the DLT evaluation period. At least 6 participants will be enrolled at the MTD/recommended phase 2 dose (RP2D).
  MTD will be evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) criteria Version 4.03
Time Frame: From first dose up to at least 28 days (Cycle 1)
Population: All treated participants
Measure: Number; unit: mg
Groups:
- Total: CC-122 administered orally on a 5 continuous days out of 7 days per week intermittent dosing schedule using active ingredient in capsule (AIC) and formulated capsules (F6)
Arm/Group | Total
Number analyzed (Participants) | 15
mg | 4.0

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study, using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) criteria version 4.03
Time Frame: From first dose to 28 days post last dose of investigational product (Up to approximately 92 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 3 | 3 | 3 | 6

4. Primary Outcome: Pharmacokinetic Parameters of CC-122: AUC0-t
Description: Area under the plasma concentration time-curve up to the last measurable concentration (AUC0-t)
Time Frame: 0, 0.5, 0.75, 1, 1.5, 3, 5, 8 and 24 hours post dose of Cycle 1 Day 1, 10, 11 or 12 (Cycle = 28 Days)
Population: Pharmacokinetics (PK) population: The PK Evaluable Population includes all participants who take at least one dose of CC- 122, and have at least one measurable CC- 122 concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*h
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
ng/mL*h
  Cycle 1 Day 1 | 634.70 (39.2) | 590.30 (6.2) | 953.89 (11.0) | 982.59 (35.9)
  Cycle 1 Day 10, 11, or 12: number analyzed (Participants) | 3 | 3 | 3 | 5
  Cycle 1 Day 10, 11, or 12 | 895.49 (45.7) | 744.65 (4.9) | 1399.3 (2.6) | 1282.80 (27.9)

5. Primary Outcome: Pharmacokinetic Parameters of CC-122: AUCtau
Description: Area under the plasma concentration time-curve during a dosing interval (AUCtau)
Time Frame: 0, 0.5, 0.75, 1, 1.5, 3, 5, 8 and 24 hours post dose of Cycle 1 Day 1, 10, 11 or 12 (Cycle = 28 Days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*h
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
ng/mL*h
  Cycle 1 Day 1 | 634.70 (39.2) | 590.3 (6.2) | 953.89 (11) | 982.59 (35.9)
  Cycle 1 Day 10, 11, or 12: number analyzed (Participants) | 3 | 3 | 3 | 5
  Cycle 1 Day 10, 11, or 12 | 895.49 (45.7) | 744.65 (4.9) | 1399.3 (2.6) | 1282.8 (27.9)

6. Primary Outcome: Pharmacokinetic Parameters of CC-122: Cmax
Description: Peak (maximum) plasma concentration (Cmax)
Time Frame: 0, 0.5, 0.75, 1, 1.5, 3, 5, 8 and 24 hours post dose of Cycle 1 Day 1, 10, 11 or 12 (Cycle = 28 Days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
ng/mL
  Cycle 1 Day 1 | 52.78 (30.4) | 52.26 (17.4) | 73.8 (20) | 107.72 (42.3)
  Cycle 1 Day 10,11 or 12: number analyzed (Participants) | 3 | 3 | 3 | 5
  Cycle 1 Day 10,11 or 12 | 72.13 (34.6) | 58.88 (28.6) | 112.61 (24.5) | 113.54 (28.7)

7. Primary Outcome: Pharmacokinetic Parameters of CC-122: Tmax
Description: Time to maximum plasma concentration (Tmax)
Time Frame: 0, 0.5, 0.75, 1, 1.5, 3, 5, 8 and 24 hours post dose of Cycle 1 Day 1, 10, 11 or 12 (Cycle = 28 Days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
hours
  Cycle 1 Day 1 | 2.24 (78.8) | 1.5 (78.5) | 1.19 (41.7) | 0.88 (46.1)
  Cycle 1 Day 10, 11 or 12: number analyzed (Participants) | 3 | 3 | 3 | 5
  Cycle 1 Day 10, 11 or 12 | 1.65 (60.1) | 1.55 (166.4) | 1.5 (78.5) | 1.28 (73.3)

8. Primary Outcome: Pharmacokinetic Parameters of CC-122: t1/2
Description: Terminal half-life of CC-122 (t1/2)
Time Frame: 0, 0.5, 0.75, 1, 1.5, 3, 5, 8 and 24 hours post dose of Cycle 1 Day 1, 10, 11 or 12 (Cycle = 28 Days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
hours
  Cycle 1 Day 1 | 11.67 (19.8) | 9.98 (19.2) | 11.67 (12.3) | 9.27 (29.9)
  Cycle 1 Day 10, 11 or 12: number analyzed (Participants) | 3 | 3 | 3 | 5
  Cycle 1 Day 10, 11 or 12 | 13.51 (28.4) | 15.5 (3) | 12.36 (11.4) | 9.7 (19.6)

9. Primary Outcome: Pharmacokinetic Parameters of CC-122: CL/F
Description: Apparent clearance (CL/F)
Time Frame: 0, 0.5, 0.75, 1, 1.5, 3, 5, 8 and 24 hours post dose of Cycle 1 Day 1, 10, 11 or 12 (Cycle = 28 Days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
L/h
  Cycle 1 Day 1 | 2.84 (35.6) | 4.11 (3.8) | 3.17 (15.8) | 2.53 (34.6)
  Cycle 1 Day 10, 11 or 12: number analyzed (Participants) | 3 | 3 | 3 | 5
  Cycle 1 Day 10, 11 or 12 | 1.55 (59.6) | 2.63 (7.5) | 2.12 (6.2) | 1.9 (30.1)

10. Primary Outcome: Pharmacokinetic Parameters of CC-122: Vz/F
Description: Apparent volume of distribution (Vz/F)
Time Frame: 0, 0.5, 0.75, 1, 1.5, 3, 5, 8 and 24 hours post dose of Cycle 1 Day 1, 10, 11 or 12 (Cycle = 28 Days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Number analyzed (Participants) | 3 | 3 | 3 | 6
L
  Cycle 1 Day 1 | 47.75 (15) | 59.11 (18.6) | 53.46 (8.5) | 33.80 (46.2)
  Cycle 1 Day 10, 11, or 12: number analyzed (Participants) | 3 | 3 | 3 | 5
  Cycle 1 Day 10, 11, or 12 | 30.29 (37.4) | 58.78 (4.5) | 37.82 (5.2) | 26.64 (31.4)

11. Primary Outcome: Accumulation Index of CC-122
Description: Accumulation Index defined as AUCtau (Cycle 1 Day 10, 11 or 12)/AUCtau (Cycle 1 Day 1)
Time Frame: 0, 0.5, 0.75, 1, 1.5, 3, 5, 8 and 24 hours post dose of Cycle 1 Day 1, 10, 11 or 12 (Cycle = 28 Days)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*h
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Number analyzed (Participants) | 3 | 3 | 3 | 5
ng/mL*h | 1.41 (9.3) | 1.26 (8.3) | 1.47 (9) | 1.25 (24.6)

12. Secondary Outcome: Best Overall Response (BOR)
Description: BOR by investigator is defined according to International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma for NHL patients and Response Evaluation Criteria in Solid Tumors (RECIST 1.1) for solid tumors patients. For NHL, complete remission (CR)=disappearance of all evidence of disease. Partial response (PR)=regression of measurable disease and no new sites. Stable disease (SD)=failure to attain CR/PR or PD. Progressive disease (PD)=any new lesion or increase by >=50% of previously sites from nadir. For solid tumors, complete response (CR)=disappearance of all target and non-target lesions and no new lesions. PR=at least a 30% decrease in the sum of diameters of target lesions and no new lesions. SD=neither sufficient shrinkage to qualify for PR or increase to qualify for PD. PD=at least 20% increase in the sum of diameters of target lesions from nadir.
Time Frame: From first dose until objectively documented progression (Up to 92 Months) at Day 15 of Cycle 2, 4, 6, and every 3 cycles thereafter (Cycle = 28 Days)
Population: Efficacy Evaluable (EE) population: all participants who complete at least one cycle of their assigned treatment regimen, and have a baseline and at least one post-baseline efficacy assessment
Measure: Count of Participants; unit: Participants
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Number analyzed (Participants) | 2 | 3 | 3 | 5
Participants
  NHL Complete Remission | 1 | 1 | 2 | 0
  NHL Partial Response (PR) | 1 | 1 | 1 | 1
  NHL Stable Disease (SD) | 0 | 1 | 0 | 2
  NHL Progressive Disease (PD) | 0 | 0 | 0 | 2
  Solid Tumors Complete Response | 0 | 0 | 0 | 0
  Solid Tumors PR | 0 | 0 | 0 | 0
  Solid Tumors SD | 0 | 0 | 0 | 0
  Solid Tumors PD | 1 | 0 | 0 | 0

13. Secondary Outcome: Duration of Response (DoR)
Description: DoR for NHL patients is defined as the time from the date when complete response (CR) or partial response (PR), whichever is first recorded are met, until the date when disease progression (PD) is first objectively documented, or the date of the last adequate tumor assessment when no disease progression is documented throughout the study according to International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma. CR=disappearance of all evidence of disease. PR=regression of measurable disease and no new sites. Progressive disease (PD)=any new lesion or increase by >=50% of previously sites from nadir.
Time Frame: as for outcome 12
Population: Efficacy Evaluable (EE) population with complete response (CR) or partial response (PR): all participants who complete at least one cycle of their assigned treatment regimen, and have a baseline and at least one post-baseline efficacy assessment
Measure: Median (Full Range); unit: weeks
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
Number analyzed (Participants) | 2 | 2 | 3 | 1
weeks | NA [24.3 to 387.0] — Median not reached as insufficient number of participants with events | NA [133.1 to 267.7] — Median not reached as insufficient number of participants with events | 139.4 [32.0 to 139.4] | 39.9 [39.9 to 39.9]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 92 months.) SAEs and Other AEs was assessed from first dose to 28 days post the last dose of study therapy (up to approximately an average of 21 months and a maximum of 92 months).
Arm/Group | AIC 2.0 mg | AIC 3.0 mg | AIC 4.0 mg | F6 3.0 mg
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 1/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/3 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIC 2.0 mg (N=3) | AIC 3.0 mg (N=3) | AIC 4.0 mg (N=3) | F6 3.0 mg (N=6)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pulmonary eosinophilia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIC 2.0 mg (N=3) | AIC 3.0 mg (N=3) | AIC 4.0 mg (N=3) | F6 3.0 mg (N=6)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 2 | 0
Eye discharge (Eye disorders) | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oedema mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 1 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 3
Thirst (General disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 3
Immunisation reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 1 | 1 | 3
Lymphocyte morphology abnormal (Investigations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 2 | 1 | 3
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 1 | 1 | 2
Urinary occult blood positive (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Mucocutaneous ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Vasospasm (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT02509039/Prot_SAP_000.pdf